CLINICAL TRIAL: NCT02234167
Title: Svenska Häktesprogrammet, Prevention, Risk Behaviour and Infectious Diseases Among IDU.
Brief Title: The Swedish Prison Program is an Intervention Prevention Program Targeting Injecting Drug Users Risk Behaviours and Infectious Diseases
Acronym: SHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Public Health Agency of Sweden (Other Government); Swedish Prison and Probation Service (Unknown); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Niklas Karlsson, PhD candidate, Karolinska Institutet
Allocation: Not Applicable | Purpose: Prevention
Other Study IDs: Swedish Prison Program
Record Dates: First submitted 2014-04-04; First posted 2014-09-09 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Having Ever Injected Drugs
MeSH Terms: interventions — Biological Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Risk behaviour and infectious diseases (Other): .(among IDU)
  Interventions: Behavioral: Risk behaviour and infectious diseases

INTERVENTIONS:
Behavioral: Risk behaviour and infectious diseases — through counselling, testing vaccination
  Other Names: biological and behavioural

SUMMARY:
The purpose of the Swedish Prison Program which started back in 1987 and up until 2009 was called "The Social Medicine Remand Prison Project" is to target injecting drug users (IDU) with primary and secondary health interventions with regards to injecting and sexual risk behaviours and infectious diseases such as hepatitis C and B, HIV and sexually transmitted infections (STI).

The overall aim is to assess the effect of different prevention efforts on HIV/HCV risk behaviour and disease outcome among IDUs over time.

DETAILED DESCRIPTION:
Risk behaviour for IDU is sexual risk taking, i.e., sex without a condom, buying or selling sex and injection risk taking, i.e., sharing needle, syringe or paraphernalia.

ELIGIBILITY:
Inclusion Criteria:

* Defined as an injecting drug user, in the prison and probation service and agree to anonymously participate

Exclusion Criteria:

* Being defined as a non-drug user, non-injecting drug user

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with injection risk behaviour | 2002-2012
  Have you received already used injection equipment from someone last 12 months Have you lent (away) already used injection equipment to someone last 12 months Have you shared solution and/or filter with someone last 12 months Number of people shared needles with last month Number of injections last month Number of Hepatitis C positive Number of HIV positive Number of Hepatitis B positive Number of respondenst positive for sexually transmitted infections

SECONDARY OUTCOMES:
Number of participants with infectious diseases | 2002-2012
  HIV, HCV, HBV and STI

CONTACTS AND LOCATIONS:
Locations (1):
- SHP, Stockholm, Sweden

REFERENCES:
- [Derived] Karlsson N, Santacatterina M, Kall K, Hagerstrand M, Wallin S, Berglund T, Ekstrom AM. Risk behaviour determinants among people who inject drugs in Stockholm, Sweden over a 10-year period, from 2002 to 2012. Harm Reduct J. 2017 Aug 16;14(1):57. doi: 10.1186/s12954-017-0184-8. PMID 28814336